CLINICAL TRIAL: NCT05354427
Title: Evaluation of Commercially Available Implantable Spacers, in Prostate Cancer Patients Undergoing Radiotherapy
Brief Title: Retrospective Evaluation of Commercial Spacers in Prostate Cancer Patients
Acronym: CLP-10095
Status: Completed | Type: Observational
Sponsor: BioProtect (Industry)
Responsible Party: Sponsor
Other Study IDs: CLP-10095
Record Dates: First submitted 2022-04-26; First posted 2022-04-29 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2022-04

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Observation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Observation — Assessment of rectal dosimetry change from pre-insertion to post-insertion in subjects with prostate cancer who have undergone radiotherapy with implantabale spacers.

SUMMARY:
Assessment of efficacy and safety of implantable spacers when used to reduce the radiation dose delivered to the organs at risk in prostate cancer patients undergoing radiotherapy.

DETAILED DESCRIPTION:
Multi-center, retrospective, observational study for assessment of rectal dose reduction following implantation of the BioProtect Balloon Implant System

ELIGIBILITY:
Inclusion Criteria:

- Males at least 18 years of age, who have undergone radiation therapy with implantable spacers

Exclusion Criteria:

* Patients whose clinical and pathological data are not available.
* Patients have been histologically diagnosed with invasive adenocarcinoma that is extracapsular with posterior extension

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Prostate Cancer
Study Population: Prostate Cancer
Sampling Method: Probability Sample
Enrollment: 175 (Actual)
Dates: Start 2020-06-18 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
Evaluation of Rectal radiation Dose | 1 month
  Dosimetry change to organs at risk in subjects with prostate cancer who have undergone radiotherapy with implantable spacers when compared to pre-implantation values.

SECONDARY OUTCOMES:
Prostate to rectum spacing | 1 month
  Measurement of prostate-rectum spacing

OTHER OUTCOMES:
Incidence of adverse events throughout the treatment course and follow up period | 3 months

CONTACTS AND LOCATIONS:
Locations (2):
- Institute of Maria Skłodowska, Curie (MCMCC), Warsaw, Poland
- Cuf Porto institution, Porto, Portugal

IPD SHARING:
Plan to Share IPD: No